CLINICAL TRIAL: NCT05187351
Title: Native Coronary Artery Instead of SAphenous Vein Graft Intervention for Treatment of Significant Saphenous Vein Graft Lesions
Status: Active, not recruiting | Type: Observational
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NASA
Record Dates: First submitted 2021-12-28; First posted 2022-01-11 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Target Vessel Failure in Saphenous Vein Grafts; Percutaneous Coronary Intervention
Keywords: Target Vessel Failure (TVF); Saphenous Vein Graft (SVG)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Percutaneous coronary intervention of the native coronary artery with Synergy — This is a registry study that will enroll patients with a 50-100% de novo SVG lesion and treated with percutaneous coronary intervention of the corresponding native coronary artery using a SYNERGY stent.

SUMMARY:
The primary study objective of the NASA registry is to evaluate the 12-month incidence of target vessel failure (TVF) in patients who present with saphenous vein graft (SVG) lesions and undergo percutaneous coronary intervention (PCI) of the corresponding native coronary artery.

DETAILED DESCRIPTION:
This is a phase IV, multi-center, single-arm, observational study evaluating the outcomes of native coronary artery PCI in patients presenting with severe SVG lesions.

Subjects will undergo clinically-indicated PCI of the native coronary artery that supplies the territory subtended by the diseased SVG at the discretion of the treating physicians.

The study team will screen and enroll patients after completion of index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Presentation with a 50-100% de novo SVG lesion that is considered to cause clinical symptoms and is treated with percutaneous coronary intervention of the corresponding native coronary artery using a SYNERGY stent.
3. Has provided informed consent and agrees to participate

Exclusion Criteria:

1. Known comorbidities/ conditions that, in the opinion of the investigator, limit life expectancy to less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a 50-100% de novo SVG lesion and treated with percutaneous coronary intervention of the corresponding native coronary artery using a SYNERGY stent.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2021-11-21 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of TVF in patients who present with SVG lesions and undergo PCI | 12 months
  Investigating the incidence of target vessel failure in patients with saphenous vein graft lesions who undergo PCI of the native coronary artery.
  or coronary bypass surgery, and tamponade requiring pericardiocentesis or surgery.

SECONDARY OUTCOMES:
Evaluate the incidence of various endpoints of patients undergoing PCI of the native coronary artery after SVG lesion development | 12 months
  The following endpoints will be measured: procedural success and complications, all cause death and cardiac death, myocardial infarction during follow up, stent thrombosis, target lesion revascularization, target vessel revascularization, non-target vessel revascularization, the composite endpoint of any death, and myocardial infarction and target vessel revascularization (patient-oriented composite endpoint), the composite endpoint of cardiac death, target vessel myocardial infarction, and target lesion revascularization (device-oriented composite endpoint for target lesion failure), and stroke.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Henry Ford Health System, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No